CLINICAL TRIAL: NCT03096080
Title: A Phase 1, Safety, Pharmacokinetic, Single Ascending Dose Study of Tesevatinib in Pediatric Subjects With Autosomal Recessive Polycystic Kidney Disease (ARPKD)
Brief Title: A Safety, Pharmacokinetic, Single Ascending Dose Study of Tesevatinib in Pediatric Subjects With Autosomal Recessive Polycystic Kidney Disease (ARPKD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kadmon Corporation, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KD019-103
Record Dates: First submitted 2017-03-06; First posted 2017-03-30 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Polycystic Kidney, Autosomal Recessive
Keywords: ARPKD; Autosomal Recessive Polycystic Kidney Disease; Pediatric Polycystic Kidney; Tesevatinib; Polycystic Kidney Disease
MeSH Terms: conditions — Polycystic Kidney, Autosomal Recessive; Polycystic Kidney Diseases | interventions — XL647

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): Single 0.25 mg/kg dose of tesevatinib
  Interventions: Drug: Tesevatinib
- Cohort 2 (Experimental): Single 0.50 mg/kg dose of tesevatinib
  Interventions: Drug: Tesevatinib
- Cohort 3 (Experimental): Single 1.00 mg/kg dose of tesevatinib
  Interventions: Drug: Tesevatinib

INTERVENTIONS:
Drug: Tesevatinib — One dose of the study drug in liquid form
  Other Names: KD019

SUMMARY:
This study evaluates safety and tolerability of a single ascending dose of a tesevatinib liquid formulation administered to pediatric subjects with ARPKD.

DETAILED DESCRIPTION:
This study is a phase 1 clinical trial focused on evaluating safety and tolerability of the Tesevatinib study drug, which is an oral solution at a 15mg/mL concentration.

To determine safety of the tesevatinib liquid formulation in pediatric subjects (age 5-12) with ARPKD, all participants receive active study drug on Day 1 of the study enrollment. To evaluate plasma pharmacokinetics (PK) of the single dose of tesevatinib in the ARPKD pediatric subjects, the blood for PK sampling is drawn on Day 1, 2, and 3 of the study. Tesevatinib dosing will be followed by a PK and a 2-week safety evaluation. After the completion of the safety review subjects may continue onto the next dosing group at the discretion of the investigator and the medical monitor.

There are three dosing arms in this study. Six participants will enroll into first dosing cohort (0.25mg/kg). Participants may be enrolled in two subsequent cohorts with increased dose (0.5mg/kg and 1.0mg/kg), if safety reporting is favorable.

Medical history will be taken at Screening Visit. Echocardiogram will be performed at Screening and Day 14. Subjects will undergo audiology testing, as well as ocular monitoring at Screening and Day 14. Blood will be drawn for a panel of laboratory tests.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of ARPKD the presence of bilaterally enlarged echogenic kidneys demonstrating poor corticomedullary differentiation and at least 1 of the following:

  1. Biliary ductal ectasia on magnetic resonance cholangiography or biliary duct ectasia or dilation on ultrasound
  2. Absence of renal cysts and/or characteristic imaging findings in both parents
  3. Signs of congenital periportal hepatic fibrosis as indicated by the presence of hepatosplenomegaly and/or esophageal varices and/or coarse liver echogenicity on ultrasound
  4. Hepatic periportal fibrosis on liver biopsy
  5. Pathologic (biopsy or autopsy) or genetic diagnosis of ARPKD in a deceased sibling or a clinical diagnosis of ARPKD in a living affected sibling
* The subject's parents or legal authorized representatives have signed a written informed consent per local regulations prior to screening. Assent, when appropriate, has been obtained from the subject according to institutional guidelines.
* The subject has a Lansky Play-Performance score of ≥ 50. Note: Subjects who are unable to walk because of paralysis, but who are in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
* The subject has the following laboratory values:

  1. Platelets > 120,000/mm3
  2. Hemoglobin > 9 g/dL
  3. Total bilirubin ≤ 1.5 mg/dL
  4. Aspartate aminotransferase (AST) < 2.5 × upper limit of normal (ULN) for age
  5. Alanine aminotransferase (ALT) < 2.5 × ULN for age
  6. eGFR ≥ 50 mL/min/1.73 m2 as measured by Chronic Kidney Disease in Children (CKiD) equation
  7. Serum potassium levels and serum magnesium levels above the lower limit of normal for age
  8. Albumin within normal limits for age
  9. Prothrombin time (PT) and partial thromboplastin time (PTT) ≤ 1.5 × ULN
* The subject has a normal ejection fraction by echocardiogram.
* The subject has a mean corrected QTcF of ≤ 450 msec.
* The subject has a blood pressure < 95th percentile for age, height, and gender. Subject may be on medication for treatment of hypertension.
* The subject has normal auditory function for age.
* If sexually active, the subject agrees to use 2 accepted methods of contraception during the course of the study and for 3 months after their last dose of study drug.

Exclusion Criteria:

* The subject has had a previous partial or total nephrectomy.
* The subject has any known genetic syndrome involving the kidney or liver other than ARPKD.
* The subject has had clinically significant gastrointestinal bleeding during the 6 months prior to enrollment.
* The subject has received any investigational therapy within 30 days prior to the first dose of study drug.
* The subject has a history of pancreatitis, has known risk factors for pancreatitis, or baseline elevations in serum amylase or lipase.
* The subject meets any of the following cardiac criteria:

  1. History of torsade de pointes, ventricular tachycardia or fibrillation, pathologic sinus bradycardia (< 50 bpm), heart block (excluding first-degree block, being PR interval prolongation only), congenital long QT syndrome or new ST segment elevation or depression or new Q wave on ECG. Subjects with a history of atrial arrhythmias should be discussed with the Medical Monitor
  2. Family history of congenital long QT syndrome or unexplained sudden cardiac death
  3. History of congenital prolonged QT syndrome, New York Heart Association class III or IV congestive heart failure
  4. History of cardiac arrhythmias, stroke, or myocardial infarction
  5. Has a cardiac pacemaker
* The subject has an abnormal baseline audiogram.
* The subject is taking or has taken any medication known to inhibit the cytochrome P450 (CYP) 3A4 isozyme or any drugs that are strong or moderate CYP3A4 inducers within 14 days prior to Day 1 of study drug.
* The subject is taking or has taken any drugs associated with torsades de pointes or known to prolong the QTc interval, including anti-arrhythmic medications within 2 weeks prior to Day 1 of study drug.
* The subject is receiving systemic anticoagulation.
* The subject has an uncontrolled intercurrent illness that would limit compliance with study requirements.
* The subject has an uncontrolled infection.
* The subject is known to be positive for the human immunodeficiency virus or hepatitis B or C.
* The subject is known to be immunocompromised.
* The subject has any medical or surgical conditions that would interfere with gastrointestinal absorption of this oral agent.
* The subject has received prior solid organ transplantation.
* The subject, in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study.
* The subject has an allergy or hypersensitivity to components of either the tesevatinib or the formulation.
* The subject is aphakic.
* The subject is pregnant or breast feeding.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2017-08-24 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Evaluation of the safety and tolerability of a single dose tesevatinib liquid formulation in pediatric participants with ARPKD | 2 weeks
  Safety and tolerability endpoints will be measured with the aggregated results of frequency and severity of adverse events and safety assessments (e.g. clinical laboratory tests, physical examinations, vital signs, ECGs, audiology testing, ocular monitoring)

SECONDARY OUTCOMES:
Evaluation of the time to peak of plasma concentration of a single dose of tesevatinib liquid formulation in pediatric participants with ARPKD. | 3 days
  Pharmacokinetic parameter Tmax for tesevatinib will be measured as time elapsed till peak concentration.
Evaluation of the plasma maximum concentration of a single dose of tesevatinib liquid formulation in pediatric participants with ARPKD. | 3 days
  Pharmacokinetic parameter Cmax for tesevatinib will be used to measure the highest concentration of the drug in plasma.
Evaluation of the Area Under the Curve (AUC) of plasma concentration against time 0-Last hours from the single dose administration of tesevatinib liquid formulation in pediatric participants with ARPKD. | 3 days
  Pharmacokinetic parameter AUC0-Last for tesevatinib will be measured and summarized by dose.
Evaluation of the Area Under the Curve (AUC) of plasma concentration against time 0-24 hours from the single dose administration of tesevatinib liquid formulation in pediatric participants with ARPKD. | 3 days
  Pharmacokinetic parameter AUC0-24 for tesevatinib will be measured and summarized by dose.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin